CLINICAL TRIAL: NCT05874986
Title: Precision Exercise (PreEx): Identifying the Determinants of Inter-individual Variation in Resistance Training Responses
Brief Title: Why do People Respond Differently to Resistance Training?
Acronym: PreEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Juha Ahtiainen, Associate Professor, University of Jyvaskyla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 60/13.00.04.00/2023
Record Dates: First submitted 2023-02-23; First posted 2023-05-25 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Exercise Training; Healthy; Skeletal Muscle Hypertrophy
MeSH Terms: interventions — Resistance Training; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (n=362) (Other): All the participants from data collection I and data collection II.
  Interventions: Other: Resistance training
- Control group (n=75) (Other): The control group consists of the participants from the training group who undergo a control period before the intervention.
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — 12-week resistance training intervention
  Other Names: Exercise training

SUMMARY:
It is well known that regular resistance training (RT) can have health benefits. However, considerable heterogeneity in RT responses has been observed. The mechanisms underlying an individual's ability to respond to RT are mainly unknown but involve a complex network of genomic and non-genomic factors. The investigators aim to examine heterogeneity in physiological responses to RT while closely monitoring other environmental factors (e.g., physical activity levels, nutrition, sleep, and stress). Participants are healthy sedentary males and females aged 18-50 (n=400). A controlled 12-week RT intervention will be conducted in two separate data collection periods due to our sample size to characterize RT response. Data will be collected before, during, and after the study period by using measurements of muscle size, physical fitness characteristics, and body composition, as well as by collecting blood samples and questionnaires. The investigators will identify the underlying factors contributing to why people differ in their physiological responses to RT. For this, comprehensive background data will be collected to identify common denominators underlying individual differences in response to RT. The investigators will use sophisticated analytical methods to reveal new predictors of training response for different traits. This research project aims to gain insight into the sources of individual variation in physiological responses to RT. On this basis, exercise training can be personalized to optimize the benefits of RT for all individuals. Ultimately, the investigators will also be able to justify better using RT as part of individualized healthcare strategies in the future.

DETAILED DESCRIPTION:
The benefits of regular resistance training (RT) are well acknowledged, but it is also well known that tremendous inter-individual variability can be detected in responses to RT. The reason(s) for individual variations in responses to RT is a very complex physiological phenomenon and is still poorly known. The individual variation in trainability suggests genetic diversity, but also non-genetic determinants potentially contribute significantly to RT responses.

The investigators hypothesize that in this study, a broad spectrum of adaptive responses to RT is detected. By scrutinizing participants' backgrounds, it can be elucidated why individuals respond differently to regular RT. Furthermore, it is hypothesized that the investigators can identify specific predictive markers for RT responsiveness. That is possible by combining information on training responsiveness with the personal characteristics of the participant.

Healthy young adults aged 18-50 will be recruited to the study in two periods to understand the biological basis of heterogeneity in RT responses by minimizing potential age and health-related physiological confounders. They are premised to respond positively to the study's primary outcome, which is the cross-sectional area (CSA) of the m. vastus lateralis (VL). To collect comprehensive data, the number of participants is maximized within the practical limitations based on our previous and extensive RT studies. Therefore, of the 400 recruited participants, 240 will first undergo 12 weeks of RT (data collection I), after which 160 participants will perform an RT period with a similar design (data collection II). Thus, an RT period will be conducted in two separate periods for both of these subsamples, as 240 is the maximum number of participants that can be supervised with our comprehensive and time-consuming physiological measures within the allocated data collection timeframe. Participants comprise an equal proportion of males and females, and sex differences in RT responsiveness will be investigated as a secondary aim of the study. Combined, data collection I and II are referred to as intervention I.

The study design of the data collection I is a single-arm trial (ethical statement number 60/13.00.04.00/2023). After assessing eligibility, participants engage in the baseline measurements and the 12-week fully supervised RT intervention. Additionally, we employ a randomized dual-trial design in data collection II (ethical statement number 1394/13.00.04.00/2023) in which one arm performs a non-RT control period before an RT period, whilst the other arm only performs RT. Moreover, test-retest baseline measurements will be performed in data collection II. The RT protocol is similar for both data collections. The participants will train two times a week, and the program will target all major muscle groups. Each training session includes exercises for the lower (leg press, knee extension) and upper body (bench press, biceps curl, and seated row). The participants will perform ~10 repetitions per set (approximately 60-80% of 1RM, 8-12 RM zone) and three working sets per exercise. The last set of each exercise is performed to momentary failure in each session. Loads are increased progressively in each exercise, session to session, during the RT period using double progression based on the final set of each exercise. A questionnaire on perceived exertion after each exercise session (sRPE) will be obtained to evaluate the participant's intrinsic effort in performing exercises. The training is executed in a local university gym with a standardized time of day, and training diaries are used to track the training loads.

The measurements are obtained at baseline and after the intervention in data collection I. Furthermore, mid-measurements are also performed in data collection II. Participants are informed of the study goals and are carefully familiarized with study protocols. All the tests are carried out at the same time of day. The participants are given feedback on their test results during the project. In addition to genetics, environmental factors are essential in explaining individuality in training responses. In this project, the investigators focus on gathering comprehensive data on variables of participants' background, nutrition, health status, and physical activity that can potentially influence the heterogeneity of RT adaptations.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* healthy (e.g., no diagnosed type 2 diabetes, cardiovascular disease, musculoskeletal disorders, etc.)
* limited experience in resistance training

Exclusion Criteria:

* medication affecting the cardiovascular system or metabolism
* metabolic, musculoskeletal, cardiovascular, or other diseases or disorders which may preclude the ability to perform exercise training and testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Change in m. vastus lateralis (VL) cross-sectional area (CSA) after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  VL CSA (cm^2) is determined at mid-thigh using a B-mode axial plane ultrasound (model SSD-α10, Aloka, Tokyo, Japan) with a 13 MHz linear-array probe (60 mm width) in extended-ﬁeld-of-view mode (23 Hz sampling frequency).
  However, since Aloka US began to show signs of malfunctioning before the onset of data collection II (approximately four months after the end of data collection I), another US device (Venue Fit R4, GE Medical Systems, USA) was used in data collection II. Due to this US-device change, test-retest measurements at baseline were performed with both devices in data collection II to enable statistical comparison of these devices later.
  GE-US was used with a L4-20t-RS linear-array probe (48,43 mm width) in extended-ﬁeld-of-view mode (6/12 MHz, 39 frames per second).

SECONDARY OUTCOMES:
Change in lower limb maximal strength after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  Maximal voluntary concentric muscle strength of leg extensors (kg) is determined in horizontal leg press device (David 210) via one-repetition maximum (1RM) test according to the NCSA guidelines. 1RM is determined with an accuracy of 2.5 kilograms.
Change in whole-body volume (cm^3) after 6 and 12-weeks of resistance training | Baseline (test and retest), week 7, week 13
  The 3D optical body (3DO) scan is used to measure whole-body volume, the volume of the body segments, and waist, hip, and thigh circumference. For 3DO, Fit3D ProScanner (Redwood City, CA, USA) is used.
Change in whole body fat-free mass after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  Fat-free body mass (kg) is measured at morning after overnight fasting by bioimpedance device (InBody 770, Biospace Co. Seoul, Korea)
Change in whole body fat mass after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  Fat body mass (kg) is measured at morning after overnight fasting by bioimpedance device (InBody 770, Biospace Co. Seoul, Korea)
Change in waist circumference after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  Waist circumference is measured by measuring tape horizontally around the waist above hipbones after exhaling in standing position
Change in grip strength after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  The maximal isometric grip strength is measured on dominant side at 90 degree elbow angle in a sitting position using a dynamometer chair (Good Strength, Metitur, Palokka, Finland)
Change in maximal vertical jump height after 6 and 12-week resistance training | Baseline (test and retest), week 7, week 13
  The countermovement jump height is calculated by measurement of flight time by jump mat
Change in blood count determined from the venous blood sample obtained at morning after overnight fasting before, and after 12-week resistance training | Baseline, week 13
  Full blood count is measured by hematology analyzer (Sysmex KX-21N, Sysmex Corp., Japan)
Change in C-reactive protein (CRP) determined from the venous blood sample obtained at morning after overnight fasting before and after 12-week resistance training | Baseline, week 13
  Serum CRP is measured by high-sensitivity ELISA kit (Quantikine HS, R&D Systems, Minneapolis, USA).
Change in metabolomics determined from the venous blood sample obtained at morning after overnight fasting before and after 12-week resistance training | Baseline, week 13
  A high-throughput serum Nuclear Magnetic Resonance (NMR) metabolomics platform will be used for the absolute quantification of serum lipids and metabolite profile.
Self-reported measure of physical activity | Baseline and after 12-weeks of RT
  Investigated by the Global Physical Activity Questionnaire (GPAQ), a standardized 16-question questionnaire that assesses categories of low, moderate, and vigorous physical activity (in MET minutes per week) in three different domains: activity at work, travel to and from places, and leisure activities. Also, sedentary behavior (minutes per week) is assessed.
Sleep self-assessment | Baseline and after 12-weeks of RT
  Investigated by The Pittsburgh Sleep Quality Index (PSQI) questionnaire which consists of questions of a four-point Likert scale (0-3), with higher scores representing greater sleep difficulties.
Self-report of eating disorder behaviors and attitudes | Baseline and after 12-weeks of RT
  Investigated by the Eating Disorder Examination Questionnaire (EDE-Q), which assesses the extent, frequency, and severity of eating disorder-related behaviors on a seven-point Likert scale or occurrence over a 28-day period. Higher scores represent higher levels of eating disorders.
Self-estimated dietary intake | Baseline and after 12-weeks of RT
  Investigated by a food frequency questionnaire (FFQ) which consists of a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period queried.
Self-estimated energy availability | Baseline and after 12-weeks of RT
  Investigated by the Low Energy Availability Questionnaire (LEAF-Q for females, LEAM-Q for men) which identifies persons at risk for low energy availability by utilizing subsets of gastrointestinal symptoms, injury frequency, and menstrual dysfunction (in women). A score ≥8 indicates that an individual is at risk for low energy availability.
Self-measure of perceived stress | Baseline and after 12-weeks of RT
  Investigated by Perceived Stress Scale (14 items); from 0 (never) to 4 (very often)

OTHER OUTCOMES:
Background information of the participants | Baseline
  Background information of the participants that are critical for training responsiveness is recorded by questionnaires, including educational and socioeconomic status (i.e., educational attainment, occupation, household income level, work and marital status, social and environmental support to exercise), history of physical training, manual labor history, medications and medical history, familial disease risks, health status (e.g. acute inflammations and acute upper respiratory infections), personality, and exercise behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Juha P Ahtiainen, Assoc.Prof., Principal Investigator — University of Jyväskylä, Faculty of Sport and Health Sciences
Locations (1):
- University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to juha.ahtiainen@jyu.fi